CLINICAL TRIAL: NCT00461955
Title: Pilot Clinical Trial of Injection of ex Vivo Amplified G-CSF Mobilised Autologous Peripheral Blood Stem Cell Transplantation in Adult Patients With Multiple Myeloma in First Response
Brief Title: Injection of ex Vivo Amplified G-CSF Mobilised Autologous Peripheral Blood Stem Cell Transplantation
Acronym: Expansion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2000/04
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Multiple Myeloma
Keywords: Symptomatic Multiple Myeloma; first line treatment; first autologous Stem Cell Transplantation; ex vivo amplified autologous peripheral blood stem cells
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): autologous peripheral blood stem cell transplantation
  Interventions: Procedure: autologous peripheral blood stem cell transplantation, ex vivo amplified

INTERVENTIONS:
Procedure: autologous peripheral blood stem cell transplantation, ex vivo amplified — autologous peripheral blood stem cell transplantation, ex vivo amplified

SUMMARY:
Hematopoietic reconstitution defined by a neutrophils number > 500/mm3 at day 7 after injection of ex vivo amplified graft and by a platelets number > 20000/mm3, at day 15 after the injection of ex vivo amplified graft, without transfusion.

DETAILED DESCRIPTION:
To check that injection of autologous peripheral blood stem cell CD34(+) "amplified ex vivo in the presence of SCF, G-CSF and TPO in HP01 Maco pharma medium culture. ": Allows to obtain a hematopoietic reconstitution:

1. Rapid : 7 days or less after the injection, regarding neutrophils and 15 days or less regarding platelets
2. Complete: numbers neutrophils and platelets respectively higher than 500/mm3 and 20000/mm3 within the times mentioned
3. Stable: no secondary neutropenia or thrombocytopenia during the year following the injection, in the absence of recurence of the myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 65 years of age
* Diagnosis of Multiple Myeloma, requiring a treatment, including high dose Melphalan whith autologous peripheral blood stem cell transplantation
* Performance status: < 2 (Karnofsky > 70%)
* Anticipated survival > 3 month
* Collection of a minimum of 10x106 cells (CD34+)/Kg of autologous G-CSF mobilised peripheral blood stem cells in 2 to 3 pheresis.
* Signed and dated informed consent

Exclusion Criteria:

* Multiple Myeloma not requiring a treatment
* Another cancer in the 5 years preceding the diagnosis or evolutive psychiatric affection
* Positive serology for HIV, hepatitis C or hepatitis B
* Hepato cellular insufficiency
* Severe renal insufficiency defined by a creatine clearance < 30 ml/mn
* Women pregnant or nursing, or effective absence of contraception
* Antecedent of serious cardiac disease in the last 6 months.
* Allergy known to the products derived from Escherichia Coli

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Hematopoietic reconstitution defined by a neutrophils number > 500/mm3 at day 7 after injection of in vitro amplified graft and by a platelets number > 20000/mm3, at day 15 after the injection of in vitro amplified graft, without transfusion. | at day 7 (neutrophils) and day 15 (platelets) after injection of in vitro amplified graft

SECONDARY OUTCOMES:
Immediate Toxicity of the injection of the amplified graft ; | just after the injection of the amplified graft
Quantitative immunological Reconstitution | at day 30, 100, 180, 270, 360 after the injection and then every 6 months
Stability of the hematopoiesis in the long term | at 1, 3, 6, 9 and 12 months after the graft
Absence of cytogenetics abnormalities not related to the multiple myeloma in the long term. | at 1, 3, 6, 9 and 12 months after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Noel MILPIED, MS, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Haut-Leveque, Pessac, France

REFERENCES:
- [Background] Bernstein ID, Andrews RG, Zsebo KM. Recombinant human stem cell factor enhances the formation of colonies by CD34+ and CD34+lin- cells, and the generation of colony-forming cell progeny from CD34+lin- cells cultured with interleukin-3, granulocyte colony-stimulating factor, or granulocyte-macrophage colony-stimulating factor. Blood. 1991 Jun 1;77(11):2316-21. PMID 1710148
- [Background] Bodine DM, Crosier PS, Clark SC. Effects of hematopoietic growth factors on the survival of primitive stem cells in liquid suspension culture. Blood. 1991 Aug 15;78(4):914-20. PMID 1714328
- [Background] Boiron JM, Marit G, Faberes C, Cony-Makhoul P, Foures C, Ferrer AM, Cristol G, Sarrat A, Girault D, Reiffers J. Collection of peripheral blood stem cells in multiple myeloma following single high-dose cyclophosphamide with and without recombinant human granulocyte-macrophage colony-stimulating factor (rhGM-CSF). Bone Marrow Transplant. 1993 Jul;12(1):49-55. PMID 8104070
- [Background] Brandt J, Srour EF, van Besien K, Briddell RA, Hoffman R. Cytokine-dependent long-term culture of highly enriched precursors of hematopoietic progenitor cells from human bone marrow. J Clin Invest. 1990 Sep;86(3):932-41. doi: 10.1172/JCI114795. PMID 1697607
- [Background] Brugger W, Heimfeld S, Berenson RJ, Mertelsmann R, Kanz L. Reconstitution of hematopoiesis after high-dose chemotherapy by autologous progenitor cells generated ex vivo. N Engl J Med. 1995 Aug 3;333(5):283-7. doi: 10.1056/NEJM199508033330503. PMID 7541111 (Retraction: PMID 11439953 Kanz L, Brugger W. N Engl J Med. 2001 Jul 5;345(1):64)
- [Background] Haylock DN, To LB, Dowse TL, Juttner CA, Simmons PJ. Ex vivo expansion and maturation of peripheral blood CD34+ cells into the myeloid lineage. Blood. 1992 Sep 15;80(6):1405-12. PMID 1381625
- [Background] Iscove NN, Shaw AR, Keller G. Net increase of pluripotential hematopoietic precursors in suspension culture in response to IL-1 and IL-3. J Immunol. 1989 Apr 1;142(7):2332-7. PMID 2784460
- [Background] Ivanovic Z, Duchez P, Dazey B, Hermitte F, Lamrissi-Garcia I, Mazurier F, Praloran V, Reiffers J, Vezon G, Boiron JM. A clinical-scale expansion of mobilized CD 34+ hematopoietic stem and progenitor cells by use of a new serum-free medium. Transfusion. 2006 Jan;46(1):126-31. doi: 10.1111/j.1537-2995.2005.00675.x. PMID 16398741
- [Background] Kobayashi M, Imamura M, Gotohda Y, Maeda S, Iwasaki H, Sakurada K, Kasai M, Hapel AJ, Miyazaki T. Synergistic effects of interleukin-1 beta and interleukin-3 on the expansion of human hematopoietic progenitor cells in liquid cultures. Blood. 1991 Oct 15;78(8):1947-53. PMID 1717075
- [Background] Moore MA. Review: Stratton Lecture 1990. Clinical implications of positive and negative hematopoietic stem cell regulators. Blood. 1991 Jul 1;78(1):1-19. No abstract available. PMID 2070044
- [Background] Moore MA. Hematopoietic reconstruction: new approaches. Clin Cancer Res. 1995 Jan;1(1):3-9. No abstract available. PMID 9815881
- [Background] Muench MO, Moore MA. Accelerated recovery of peripheral blood cell counts in mice transplanted with in vitro cytokine-expanded hematopoietic progenitors. Exp Hematol. 1992 Jun;20(5):611-8. PMID 1587307
- [Background] Muench MO, Schneider JG, Moore MA. Interactions among colony-stimulating factors, IL-1 beta, IL-6, and kit-ligand in the regulation of primitive murine hematopoietic cells. Exp Hematol. 1992 Mar;20(3):339-49. PMID 1373685
- [Background] Reiffers J, Marit G, Vezon G, Cony-Makhoul P, Boiron JM, Montastruc M, Rice A, Broustet A. Autologous blood stem cell grafting in hematological malignancies. Present status and future directions. Transfus Sci. 1992;13(4):399-405. doi: 10.1016/0955-3886(92)90024-B. No abstract available. PMID 10147738
- [Background] Reiffers J, Faberes C, Boiron JM, Marit G, Foures C, Ferrer AM, Cony-Makhoul P, Puntous M, Bernard P, Vezon G, et al. Peripheral blood progenitor cell transplantation in 118 patients with hematological malignancies: analysis of factors affecting the rate of engraftment. J Hematother. 1994 Fall;3(3):185-91. doi: 10.1089/scd.1.1994.3.185. PMID 7530133
- [Background] Rice A, Boiron JM, Barbot C, Dupouy M, Dubsoc-Marchenay N, Dumain P, Lacombe F, Reiffers J. Cytokine-mediated expansion of 5-FU resistant peripheral blood stem cells and bone marrow: self-renewal and commitment capacity. J Hematother. 1994 Summer;3(2):135-9. doi: 10.1089/scd.1.1994.3.135. PMID 7522897
- [Background] Shih JP, Ogawa M. Monoclonal antibody J11d.2 recognizes cell cycle-dormant, primitive hematopoietic progenitors of mice. Blood. 1993 Mar 1;81(5):1155-60. PMID 8443377
- [Background] Smith C, Gasparetto C, Collins N, Gillio A, Muench MO, O'Reilly RJ, Moore MA. Purification and partial characterization of a human hematopoietic precursor population. Blood. 1991 May 15;77(10):2122-8. PMID 1709369